CLINICAL TRIAL: NCT00173277
Title: Screening for CRC Using a Mixed Strategy of Sigmoidoscopy and Colonoscopy in Average-Risk Population According to Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700610
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
BACKGROUND: Primary screening with sigmoidoscopy would miss a substantial proportion of advanced proximal neoplasia (APN), but screening with universal colonoscopy is costly. The aim of this study is to assess the efficacy of mixed strategy which uses sigmoidoscopy for younger patients and colonoscopy for older patients.

MATERIALS and METHODS: We analyzed an established database containing consecutive average-risk adults aged 50 or older who underwent screening colonoscopy as part of health check-up. We assessed the efficacy of mixed screening strategy using colonoscopy for persons aged at and above a certain cut-off age and sigmoidoscopy for persons aged below that age. Those who underwent sigmoidoscopy initially would be referred for subsequent colonoscopy if distal sentinel lesion was detected.

DETAILED DESCRIPTION:
Because the prevalence of proximal colon cancer and APN was higher in older patients15, a greater proportion of advanced colonic neoplasia or cancer would be missed if colonoscopy was not performed for older patients. So if we develop a mixed strategy to offer sigmoidoscopy for younger patients and reserve colonoscopy for older patients, we might be able to detect more APN with fewer colonoscopic procedures. We aimed to determine an optimal cut-off age and choose an appropriate distal sentinel lesion for subsequent colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Only asymptomatic ethnic Chinese subjects aged 50 years or older who underwent total colonoscopy were included in this study

Exclusion Criteria:

* Persons with symptoms indicative of colorectal cancer, such as hematochezia, body weight loss, development of persistent abdominal pain or rectal pain, and a change in bowel habit, were excluded from this study. Other exclusion criteria were: (1) past history of CRC, colon polyps, or inflammatory bowel disease; (2) a history of screening tests, including FOBT, sigmoidoscopy, colonoscopy, or barium studies within 5 years; (3) any first degree relative(s) with colon cancer; (4) criteria for hereditary nonpolyposis colorectal cancer, familial adenomatous polyposis, or other polyposis syndrome; (5) obvious anemia with hemoglobin level less than 10g/dl; (6) incomplete examination of entire colon, including poor colon preparation and failure to reach cecum.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500
Dates: Start 2003-06; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Study Director — Departments of Internal Medicine, National Taiwan University Hospital, National Taiwan University College of Medicine, Taipei, Taiwan
Locations (1):
- Departments of Internal Medicine, Medicine National Taiwan University Hospital,, Taipei, Taiwan

REFERENCES:
- [Background] Lieberman DA, Weiss DG, Bond JH, Ahnen DJ, Garewal H, Chejfec G. Use of colonoscopy to screen asymptomatic adults for colorectal cancer. Veterans Affairs Cooperative Study Group 380. N Engl J Med. 2000 Jul 20;343(3):162-8. doi: 10.1056/NEJM200007203430301. PMID 10900274